CLINICAL TRIAL: NCT02645760
Title: Comparison of Core Stabilization Exercise and Physical Therapy Treatment in Patients With Subacute Non-specific Low Back Pain
Brief Title: Effectiveness of Core Stabilization Exercise in Patients With Subacute Non-Specific Low Back Pain
Acronym: CSENSLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Rungthip Chalermsan, Faculty of Associated Medical Sciences, Khon Kaen University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KKU-571H106
Record Dates: First submitted 2015-12-31; First posted 2016-01-05 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2015-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core stabilization exercise (Active Comparator): 7-weeks of core stabilization exercise
  Interventions: Other: Core stabilization exercise
- conventional treatment (Active Comparator): 7-weeks of conventional treatment include therapeutic ultrasound and hot pack
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Core stabilization exercise — 7-weeks of core stabilization exercise
  Arms: Core stabilization exercise
Other: Conventional treatment — 7-weeks of conventional treatment include therapeutic ultrasound and hot pack
  Arms: conventional treatment

SUMMARY:
The purpose of this study is to examines the effectiveness of Core stabilization exercise on pain intensity at rest, functional disability, lumbar movement and ability to perform repositioning tasks (joint position sense) in patients with subacute non-specific low back pain.

DETAILED DESCRIPTION:
This study is to compare the effectiveness of Core stabilization exercise and physical therapy on pain intensity at rest, functional disability, lumbar movement and ability to perform repositioning tasks (joint position sense) in patients with subacute non-specific low back pain. There are 2 groups receiving 2 different kinds of intervention: treatment group receiving core stabilization exercise (CSE) and control group receiving physical therapy including therapeutic ultrasound and hydrocollator pack. Each intervention will perform for 7 weeks. The patients will assess for all outcome measures at baseline, 7 weeks of intervention, and 1- month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Onset of back pain within 6 -12 weeks participants had no history of back pain for a period of 6 months prior to the current episode.
* Pain intensity measure by a numerical rating scale (0-10 NRS) and a score of pain at least 3 out of 10.
* Never receive the treatment by core stabilization exercise (CSE) during 3 months before participate in this study.

Exclusion Criteria:

* Pregnancy
* Onset of serious spinal pathology: spinal fracture, spinal tumor or spinal infection.
* Cauda equina syndrome.
* Presented at least 2 out of 3 signs of neurological deficit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rungthip Chalermsan, Study Director — Faculty of Associated Medical Sciences, Khon Kaen University
Locations (1):
- Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Stabilization Exercise: 7-weeks of core stabilization exercise Participants were received treatment with Core stabilization exercise (CSE) which applied from the treatment approaches of Puntumetakul et al (2013). 20-minute sessions, 2 sessions per week all over 7 weeks by a physical therapist (researcher number 2) and home exercises every day with recording this practice (duration and frequency of exercise) in the diary over the study period. This exercise aims for training the activation of the local muscle system (the deep muscle layer) in
- Conventional Treatment: 7-weeks of conventional treatment include therapeutic ultrasound and hot pack Participants were received 5 minutes of therapeutic ultrasound which used a 1-MHz ultrasound frequency with the intensity of 0.8-1.0 W/cm2 by continuous mode. The sound head moved in small circles or longitudinal strokes around the painful area of lower back in a side lying position. The participant was received 15 minutes of the hydrocollator pack therapy (60 °C) which placed under the painful area of lower back in a supine lying position after receive therapeutic ultrasound.
Period: Overall Study
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data was presented as means, standard deviations (SD) and 95% CI. The statistical analysis performed using SPSS version 16.0 for windows (IBM Corporation, Armonk, NY, USA). The Shapiro-Wilk used to test for the normality of the data.
Groups:
- Core Stabilization Exercise: 7-weeks of core stabilization exercise Participants were received treatment with Core stabilization exercise (CSE) which applied from the treatment approaches of Puntumetakul et al (2013). 20-minute sessions, 2 sessions per week all over 7 weeks by a physical therapist (researcher number 2) and home exercises every day with recording this practice (duration and frequency of exercise) in the diary over the study period. This exercise aims for training the activation of the local muscle system (the deep muscle layer) including the transversus abdominis (TrA) and lumbar multifidus (LM) muscles.
- Total: Total of all reporting groups
Arm/Group | Core Stabilization Exercise | Conventional Treatment | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.63 (10.26) | 37.89 (10.60) | 38.76 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 3 | 1 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.97 (3.07) | 24.03 (4.08) | 24.50 (3.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain on 11- Point Numerical Rating Scale at Week 7
Description: The 11 point numerical rating scale (11-NRS) is a method to measure pain intensity. The zero represents no pain while 10 represent the worst imaginable pain.The patient is asked to cross or circle a score that the best represents the pain intensity. Change = (week 7 score - baseline score)
Time Frame: baseline an week 7
Population: Analysis of covariance (ANCOVA) was performed to compare differences between groups for outcome measures. To estimate the adjusted mean differences and the 95% confidence intervals for each outcome measure of each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Number analyzed (Participants) | 19 | 19
units on a scale | 1.32 (1.83) | 3.63 (1.64)
Statistical Analysis 1: Comparison: Core Stabilization Exercise vs Conventional Treatment; It was calculated that 38 participants randomized in a 1:1 fashion between the 2 arms would have at least 80% power to detect a difference of 2.26 points in mean 11-point NRS pain score between core stabilization exercise and conventional treatment from baseline to week 7; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in Functional Disability on Roland-Morris Disability Questionnaire at Week 7
Description: This outcome was assessed by the Roland-Morris disability questionnaire (RMDQ) Thai version that is designed to assess self-rated physical disability caused by LBP. This questionnaire has 24 items. The participant put a tick on the statement when it applies to him that specific day. The scores range from 0 (no disability) to 24 (maximum disability). change = (baseline score - week 7 score
Time Frame: baseline and week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Number analyzed (Participants) | 19 | 19
units on a scale | 1.53 (2.29) | 4.89 (4.18)
Statistical Analysis 1: Comparison: Core Stabilization Exercise vs Conventional Treatment; It was calculated that 38 participants randomized in a 1:1 fashion between the 2 arms would have at least 80% power to detect a difference of 2.68 points in mean disability score (RMDQ score) between core stabilization exercise and conventional treatment from baseline to week 7; Test type: Superiority or Other; p = 0.009, ANCOVA

3. Secondary Outcome: Change From Baseline in Back Range of Motion (Flexion) on Modified-modified Schober's Test at Week 7
Description: Modified-modified Schober's test used a tape measure held directly over the spine between points 15 cm above the posterior superior iliac spine (PSIS) with the participant in the neutral standing position on the foot print. The participant was asked to stand with knees locked and bend forward (lumbar flexion) as far as possible without pain; the increase in distance between the marks gave an estimate of lumbar ROM. change =(baseline score - week 7 score)
Time Frame: baseline and week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Number analyzed (Participants) | 19 | 19
centimeter | 5.32 (1.51) | 4.32 (0.73)
Statistical Analysis 1: Comparison: Core Stabilization Exercise vs Conventional Treatment; It was calculated that 38 participants randomized in a 1:1 fashion between the 2 arms would have at least 80% power to detect a difference of 0.79 centimeter in mean range of motion between core stabilization exercise and conventional treatment from baseline to week 7; Test type: Superiority or Other; p = 0.013, ANCOVA

4. Secondary Outcome: Change From Baseline in Repositioning Error on Repositioning Test at Week 7
Description: This test was performed by measuring how accurately the participant during sitting that could reposition the lumbar spine into the former lumbar position, after change position in the sagittal plane. The procedure use a laser pointer adjusted to be level, was positioned to have the mark line directly on 0 cm. After having actively moved around, in maximum flexion-extension and return to neutral position, the laser line on the tape-measure, the deviation from the 0 point was measured in centimeter. change = (baseline score - week 7 score)
Time Frame: baseline and week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Number analyzed (Participants) | 19 | 19
centimeter | 0.43 (0.34) | 0.67 (0.42)
Statistical Analysis 1: Comparison: Core Stabilization Exercise vs Conventional Treatment; It was calculated that 38 participants randomized in a 1:1 fashion between the 2 arms would have at least 80% power to detect a difference of 0.30 centimeter in mean repositioning error between core stabilization exercise and conventional treatment from baseline to week 7; Test type: Superiority or Other; p = 0.012, ANCOVA

ADVERSE EVENTS:
Arm/Group | Core Stabilization Exercise | Conventional Treatment
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes